CLINICAL TRIAL: NCT02816164
Title: A Multi Centre Study to Compare Administration Schedules of G-CSF (Filgrastim) for Primary Prophylaxis of Chemotherapy-Induced Febrile Neutropenia in Early Stage Breast Cancer (REaCT-G2)
Brief Title: A Study to Compare Administration Schedules of G-CSF (Filgrastim) for Primary Prophylaxis of Febrile Neutropenia
Acronym: REaCT-G2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTT 16-04
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Early Stage Breast Cancer
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neupogen for 5 days (Active Comparator): Neupogen injection for 5 days
  Interventions: Drug: Neupogen
- Neupogen for 7 days (Active Comparator): Neupogen injection for 7 days
  Interventions: Drug: Neupogen
- Neupogen for 10 days (Active Comparator): Neupogen injection for 10 days
  Interventions: Drug: Neupogen

INTERVENTIONS:
Drug: Neupogen — Subcutaneous injections
  Other Names: Filgrastim

SUMMARY:
In patients with early-stage breast cancer, chemotherapy has substantially improved survival rates. Improvements in outcomes, however, are compromised by the considerable toxicities associated with chemotherapy, the most notable being neutropenia. Neutropenia is the presence of abnormally few white blood cells, leading to increase susceptibility to infection and can require hospitalization and need for intravenous antibiotics and is sometimes fatal. Febrile neutropenia (FN) can also be associated with treatment delays and dose reductions, potentially compromising treatment efficacy. Patients can receive medication to reduce the risk of FN such as Neupogen (filgrastim) as a daily injection for 5, 7 or 10 days. Since there is genuine uncertainty among healthcare professionals as to which administration schedule of Neupogen is the best for patients, the investigators are performing a randomized study for which patients will receive either 5, 7 or 10 days of Neupogen. Neupogen can cost approximately $200/injection, so if a physician prescribes 10 days for 8 cycles of treatment, this can cost $16,000 compared to a 5 day treatment which would cost half this. In addition to cost savings, many patients are not able to give themselves injections on a daily basis and require nursing resources which are utilized at high cost. This study will use an oral consent model to compare 5, 7 and 10 days of Neupogen to evaluate rates of febrile neutropenia and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer
* Planned to start docetaxel component of FEC-D or AC-D, or first cycle of; dose-dense AC-T, TC, FEC-D or TAC chemotherapy
* ≥19 years of age
* Able to provide verbal consent

Exclusion Criteria:

* Contraindication to Filgrastim

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Febrile neutropenia | 2 years
  Number of participants with febrile neutropenia
Treatment-related hospitalization | 2 years
  Number of participants admitted to emergency for treatment-related reasons

SECONDARY OUTCOMES:
Chemotherapy dose delay | 2 years
  Number of participants who experience a dose delay with their chemotherapy treatment
Chemotherapy dose reduction | 2 years
  Number of participants who experience a dose reduction in their chemotherapy treatment
Chemotherapy discontinuation | 2 years
  Number of participants who stop chemotherapy for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Derived] Clemons M, Fergusson D, Simos D, Mates M, Robinson A, Califaretti N, Zibdawi L, Bahl M, Raphael J, Ibrahim MFK, Fernandes R, Pitre L, Aseyev O, Stober C, Vandermeer L, Saunders D, Hutton B, Mallick R, Pond GR, Awan A, Hilton J. A multicentre, randomised trial comparing schedules of G-CSF (filgrastim) administration for primary prophylaxis of chemotherapy-induced febrile neutropenia in early stage breast cancer. Ann Oncol. 2020 Jul;31(7):951-957. doi: 10.1016/j.annonc.2020.04.005. Epub 2020 Apr 20. PMID 32325257